CLINICAL TRIAL: NCT04639921
Title: Non Celiac Gluten Sensitivity, a Double Blind Placebo Controlled Food Challenge With Cross-over in Healthy Danish Adolescents
Brief Title: Non Celiac Gluten Sensitivity, DBPCFC in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Steffen Husby, MD, Professor, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OUH-HCA 004
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Non-celiac Gluten Sensitivity; Adolescents

STUDY DESIGN:
Intervention Model Description: Diagnostic double blind randomized placebo controlled food challenge with cross over
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind performed by food provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active - placebo (Experimental): intake of socalled gluten bars two daily for seven days, followed by one week wash-out, and then placebo bars for seven days
  Interventions: Diagnostic Test: positive test followed by gluten-free diet; Dietary Supplement: Placebo
- placebo - active (Placebo Comparator): intake of placebo bars two daily, followoed by wash-out for one week, and gluten bars (experimental) for seven days.
  Interventions: Diagnostic Test: positive test followed by gluten-free diet; Dietary Supplement: Placebo

INTERVENTIONS:
Diagnostic Test: positive test followed by gluten-free diet — DBPCFC with gluten
Dietary Supplement: Placebo — Placebo

SUMMARY:
In a population based on healthy adolescents we will conduct a double blind placebo controlled food challenge (DBPCFC) with cross-over to identify patients with NCGS as recommended by the socalled Salerno criteria. It will take place at Hans Christian Andersen Childrens Hospital at Odense University Hospital, Denmark in October-November 2020.

DETAILED DESCRIPTION:
Non Gluten Sensitivity, a double blind placebo controlled food challenge with cross-over in healthy Danish Adolescents

Caecilie Crawley, Nadia Savino, Cecilie Halby, Stine Dydensborg Sander, Anne-Marie Nybo Andersen, Joseph Murray, Robin Christensen, Steffen Husby

INTRODUCTION Non-celiac gluten sensitivity (NCGS) is a newly described disease entity, where the individual shows signs of sensitivity to gluten, but with no evidence of IgE-mediated wheat allergy or CD (1). The extent and severity of NCGS is so far an enigma (2), but symptoms of NCGS may be commonly occurring, with a reported prevalence of up to 6% of the adult population (3). So far, only ten studies with a double-blind placebo-controlled food challenge have been performed showing divergent study outcomes due to different study designs and methods and a significant nocebo/placebo effect. In general, the studies are characterized by patient recruitment from a gastroenterological clinic limited to adults (4). Our study stands out in this respect, as we will investigate an unselected group of patients as adolescents (not recruited from an outpatient clinic), because patients with NCGS often report that their symptoms started at that time.

Several researchers have concluded that patients with NCGS may not react to gluten but instead to dietary carbohydrates, so-called FODMAPS or amylase trypsin inhibitors (5). A study with Double Blind Placebo Controlled Food Challenges by Lundin et al. (6) has been published but with inconclusive results. Given this background, contrary to CD, factors involved in the etiology of NCGS are still unknown. In a search for biomarkers and perhaps even contributing factors for NCGS, a microbial signature of the gut would be a good candidate.

METHODS Study Design In a population based on healthy adolescents we conducted a double blind placebo controlled food challenge (DBPCFC) with cross-over to identify patients with NCGS as recommended by the Salerno criteria(1). It will take place at Hans Christian Andersen Childrens Hospital at Odense University Hospital, Denmark in November 2020. It was approved by The Regional Committees on Health Research Ethics for Southern Denmark (project no S-20160061) and the Danish Protection Agency (2008-58-0018).

Study Population The adolescents were participants in the GlutenFunen cohort, which were recruited from an unselected subsample of the Danish National Birth Cohort, defined as those living on the Island of Funen, Denmark. The Danish National Birth Cohort consists of approx. 96,000 children, who are followed from intrauterine life and onwards (most recent follow-up is 18-years follow-up)(7). Their mothers were recruited from 1996 to 2002 from the general population with a participation rate of approximately 30%.

The GlutenFunen cohort included 1266 out of the 7431 eligible participants (17%), in the age 15-21 years old and were examined for Coeliac Disease, anthropometric and metabolic measurements. Furthermore, the participants in the GlutenFunen cohort answered a questionnaire about their gastrointestinal symptoms, and a score based on the number of gastrointestinal symptoms was calculated. Criteria for inclusion was a score higher than three, in total 273 participants. They were all contacted by phone by the author NS or CC and invited to an information meeting where a dietician instructed how to follow a gluten free diet.

Exclusion criteria were wheat allergy, transglutaminase IgA higher than reference range, Inflammatory Bowel Disease and current antibiotic treatment Study Intervention The study was arranged in two phases. See figure 1. The first phase began with a run-in period of seven days to adapt the gluten free diet, subsequent one week of gluten free diet. If the participants responded to the gluten free diet defined as a VAS score higher than 25% compared to initial VAS score the participants proceeded to phase two.

Phase two consisted of three periods each lasting seven days; The first being a challenge with gluten/placebo, then a wash-out phase, and finally the second challenge with placebo/gluten. During the whole study, the participants had to follow a strict gluten free diet. Adherence was not evaluated during the trial, but the participants were asked to note whether they accidentally had eaten gluten.

The granola bars The participants had to eat two granola bars every day except for the wash-out period. The granola bar was lactose free and low in FODMAPS and the amount of gluten in the gluten containing granola bar was 5.0g. The recipe was kindly provided by Lundin et al. (6). In a triangle test there were no difference regarding taste, look and consistency between the gluten and the placebo granola bar.

Outcome measures Gastrointestinal symptoms were measured with a self-administrated 10 items questionnaire, which represented a modified gastrointestinal symptom rating score. It was assessed on a 100mm visual analog scale (VAS) (1-100) at day 1 and 13 and day 15-35. A total score was calculated as the mean of the 10 items. Extraintestinal symptoms and mental health symptoms were measured with SF-36 and the Warwick-Edinburgh Mental well-being scale (14 items) at day 1, 14, 21, 28 and 35.

The Microbiome The participants had to deliver a faecal sample at day 1, 14, 21,28 and 35. To ensure a high compliance the faecal sample was collected at the home of the participants. The faecal sample was frozen immediately, as described previously (8).

Randomization and blinding. The participants were randomised to placebo-gluten or gluten-placebo in blocks of four by the randomization module in RedCap administrated by the data-manager of the study. The kitchen of Odense University Hospital baked the granola bars and packed them in different boxes with two colours to ensure the blinding of the study for the investigators and the participants. The randomization code was not revealed before the end of the trial.

Outcome The primary outcome was identifying participants with NCGS defined as a 30% worsening of symptoms when eating gluten compared to the placebo based on the modified VAS score.

The secondary outcome was an improvement in the mental health of the participants when living on the gluten free diet.

The tertiary outcome was to identify microbial signatures in patients with NCGS.

Statistical analysis Normally distributed data were described with means and the standard deviation and they were compared using paired t-test. Non-parametric data were described with median and percentiles and compared using Mank-Whitney Rank sum test ??. P-values < 0.05 was considered significant.

Power Assuming a positivity of 30% to the challenge, a power of 80% and a significance level of 5% we calculated a need for 29 participants.

ELIGIBILITY:
Inclusion Criteria:

* positive questionnaire of at least 3 predefined symptoms, from cohort study

Exclusion Criteria:

* not 3 predefined symptoms, from cohort study

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
symptom VAS score | one week
  score from 0-100

SECONDARY OUTCOMES:
specific symptoms | one week
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Husby, M.D., Study Director — Odense University Hospital
Locations (1):
- Steffen Husby, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available in a pseudo-anonymized form to researchers from the Danish National Cohort
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2021-2026
Access Criteria: Researchers from the Danish National Birth Cohort

REFERENCES:
- [Result] Catassi C, Elli L, Bonaz B, Bouma G, Carroccio A, Castillejo G, Cellier C, Cristofori F, de Magistris L, Dolinsek J, Dieterich W, Francavilla R, Hadjivassiliou M, Holtmeier W, Korner U, Leffler DA, Lundin KE, Mazzarella G, Mulder CJ, Pellegrini N, Rostami K, Sanders D, Skodje GI, Schuppan D, Ullrich R, Volta U, Williams M, Zevallos VF, Zopf Y, Fasano A. Diagnosis of Non-Celiac Gluten Sensitivity (NCGS): The Salerno Experts' Criteria. Nutrients. 2015 Jun 18;7(6):4966-77. doi: 10.3390/nu7064966. PMID 26096570
- [Result] Husby S, Murray J. Non-celiac gluten hypersensitivity: What is all the fuss about? F1000Prime Rep. 2015 May 12;7:54. doi: 10.12703/P7-54. eCollection 2015. PMID 26097727
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Francavilla R, Cristofori F, Castellaneta S, Polloni C, Albano V, Dellatte S, Indrio F, Cavallo L, Catassi C. Clinical, serologic, and histologic features of gluten sensitivity in children. J Pediatr. 2014 Mar;164(3):463-7.e1. doi: 10.1016/j.jpeds.2013.10.007. Epub 2013 Nov 16. PMID 24252792
- [Result] Biesiekierski JR, Newnham ED, Shepherd SJ, Muir JG, Gibson PR. Characterization of Adults With a Self-Diagnosis of Nonceliac Gluten Sensitivity. Nutr Clin Pract. 2014 Aug;29(4):504-509. doi: 10.1177/0884533614529163. Epub 2014 Apr 16. PMID 24740495
- [Result] Skodje GI, Sarna VK, Minelle IH, Rolfsen KL, Muir JG, Gibson PR, Veierod MB, Henriksen C, Lundin KEA. Fructan, Rather Than Gluten, Induces Symptoms in Patients With Self-Reported Non-Celiac Gluten Sensitivity. Gastroenterology. 2018 Feb;154(3):529-539.e2. doi: 10.1053/j.gastro.2017.10.040. Epub 2017 Nov 2. PMID 29102613
- [Result] Olsen J, Melbye M, Olsen SF, Sorensen TI, Aaby P, Andersen AM, Taxbol D, Hansen KD, Juhl M, Schow TB, Sorensen HT, Andresen J, Mortensen EL, Olesen AW, Sondergaard C. The Danish National Birth Cohort--its background, structure and aim. Scand J Public Health. 2001 Dec;29(4):300-7. doi: 10.1177/14034948010290040201. PMID 11775787
- [Result] Kyhl HB, Jensen TK, Barington T, Buhl S, Norberg LA, Jorgensen JS, Jensen DF, Christesen HT, Lamont RF, Husby S. The Odense Child Cohort: aims, design, and cohort profile. Paediatr Perinat Epidemiol. 2015 May;29(3):250-8. doi: 10.1111/ppe.12183. Epub 2015 Mar 10. PMID 25756293
- [Derived] Crawley C, Savino N, Halby C, Sander SD, Andersen AN, Arumugam M, Murray J, Christensen R, Husby S. The effect of gluten in adolescents and young adults with gastrointestinal symptoms: a blinded randomised cross-over trial. Aliment Pharmacol Ther. 2022 May;55(9):1116-1127. doi: 10.1111/apt.16914. Epub 2022 Mar 29. PMID 35352373